CLINICAL TRIAL: NCT06147466
Title: Time Spent In the Target Glucose Range and MatErnaL and Neonatal Effects in Women With tYpe 2 Diabetes in Pregnancy (TIMELY)
Brief Title: Time Spent In Target Glucose Range in Women With T2D Diabetes in Pregnancy
Acronym: Timely
Status: Recruiting | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: University of Manitoba (Other); Women's College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 21-0065-E
Record Dates: First submitted 2023-04-03; First posted 2023-11-27 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-03

CONDITIONS: Diabete Type 2; Pregnancy in Diabetic
Keywords: glucose range; neonatal outcomes; glycemic control; hypoglycemia; insulin resistance; preganant; pregnancy; CGM; Continuous Glucose Monitoring; Dexcom; maternal outcomes; Pregnancy in Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pregnancy in Diabetics; Hypoglycemia; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Dexcom Continuous Glucose Monitoring — A continuous glucose monitor (CGM) is a wearable device that tracks blood glucose (sugar) every few minutes, throughout the day and night. The readings are relayed in real time to a device which can be read by the patient, caregiver or health-care provider, even remotely

SUMMARY:
Prospective cohort study to determine to what extent women with type 2 diabetes are achieving the time in the target range outlined for women with type 1 diabetes (70-140 mg/dl or 3.5-7.8 mmol/l), overall and by trimester, by standard CGM measures and functional data analysis

ELIGIBILITY:
Inclusion Criteria:

1. Women with type 2 diabetes diagnosed prior to pregnancy or prior to 20 weeks gestation with either a HbA1c of >6.5%, fasting glucose ≥7.0, or 2 hr glucose ≥11.1 on a 75g OGTT. To make the diagnosis in pregnancy one needs 2 values equal to or greater than the values above.
2. ≤14 weeks gestation,
3. age ≥18 years
4. Willingness to use the study devices a minimum of 10 days per trimester
5. Able to provide informed consent
6. Have access to email

Exclusion Criteria:

1. Non-type 2 diabetes
2. Current treatment with drugs known to interfere with glucose metabolism as judged by the investigator such as high dose systemic corticosteroids
3. Known or suspected allergy against insulin
4. Women with nephropathy (eGFR<30), severe autonomic neuropathy, uncontrolled gastroparesis that, as judged by the investigator, is likely to interfere with the normal conduct of the study and interpretation of study results
5. Severe visual or hearing impairment, as judged by the investigator to impact treatment compliance
6. Unable to communicate effectively in English as judged by the investigator
7. Any reason judged by the investigator that would likely interfere with the normal conduct of the study and interpretation of study results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant Women with Type 2 diabetes with either a HbA1c of >6.5%, fasting glucose ≥7.0, or 2 hr glucose ≥11.1 on a 75g OGTT
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Time in target range | 7-9 months
  To determine to what extent women with type 2 diabetes are achieving the time in the target range outlined for women with type 1 diabetes (70-140 mg/dl or 3.5-7.8 mmol/l), overall and by trimester, by standard CGM measures and functional data analysis

SECONDARY OUTCOMES:
Delivery outcome | 7-9 months
  delivery outcome will be reported as ,full term birth, pre-term birth, spontaneous abortion, miscarriage or termination.
Maternal outcome | 7-9 months
  Date and time of hospital admission for delivery and discharge.
Maternal outcome (HTN) | 7-9 months
  Maternal postpartum diagnosis of hypertension or pre-eclampsia.
Neonatal weight at birth | 7-9 months (Delivery of neonate)
  Neonatal weight measurement collected from medical chart.
Neonatal outcomes (hypoglycemia) | 7-9 months (Delivery of neonate)
  Proportion of babies born with hypoglycemia. The lowest recorded glucose value (mmol/L) will be collected for babies born with hypoglycemia
Neonatal outcomes (chromosomal abnormality) | 7-9 months (Delivery of neonate)
  Proportion of babies born with chromosomal abnormality and type of chromosomal abnormality
Neonatal outcomes (congenital anomaly) | 7-9 months (Delivery of neonate)
  Proportion of babies born with congenital anomaly and type of congenital anomaly
Neonatal outcomes (birth injury) | 7-9 months (Delivery of neonate)
  Proportion of babies born with neonatal birth injury and type of injury
Neonatal outcomes (hyperbilirubinemia) | 7-9 months (Delivery of neonate)
  Proportion of babies born with neonatal hyperbilirubinemia requiring treatment (• phototherapy > 6 continuous hours, an exchange transfusion, intravenous gamma globulin or required re-admission into hospital during the first 7 days of life)
Neonatal outcomes (neonatal intensive care admission) | Delivery of neonate to 6 weeks postpartum
  Proportion of babies admitted to neonatal intensive care admission
Covariates (maternal obesity) | 16-24 weeks gestation, 34 weeks gestation, 4-6 weeks postpartum
  maternal weight will be collected/measured
Covariates (maternal ethnicity) | Enrollment (16-24 weeks gestation)
  maternal ethnicity will be collected
Covariates (Mother's total household income) | enrollment 16-24 weeks gestation
  total household income will be collected
Adverse events | 7-9 months
  Adverse events description and time of occurrence will be recorded when applicable
Blood Insulin | at 16-24 weeks gestation
  blood insulin measured in pmol/L.
Measures of insulin resistance (HOMA-IR ) | at 16-24 weeks gestation
  Homeostatic Model Assessment for Insulin Resistance ( HOMA-IR ) index will be calculated suing blood insulin and blood glucose
Mean blood glucose measurement | at 16-24 weeks gestation
  Blood glucose measured in mmol/L
Diabetes distress | at 16-24 weeks gestation and at 34 weeks gestation
  Using Diabetes Distress Screening Scale (DDSS17). The scale yields an overall distress score based on the average of response on the 1-6 scale for all 18 items. The DDS-17 identifies three levels of specificity of diabetes distress information for use in clinical care, from overall emotional distress related to diabetes to highly specific sources of diabetes distress. Higher score is worse.
Sleep quality | at 16-24 weeks gestation and at 34 weeks gestation
  Using the Berlin Questionnaire. The Berlin Questionnaire consists of three categories designed to elicit information regarding snoring (category 1), daytime somnolence (category 2), and the presence of obesity and/or hypertension (category 3). Categories 1 and 2 are considered positive if 2 or more responses are positive category 3 is considered positive if 1 response is positive and/or the body mass index is greater than 30 kg per meter squared. A patient is considered to have a high likelihood of sleep disordered breathing if 2 or more categories are positive
Sleep apnea | at 16-24 weeks gestation and at 34 weeks gestation
  Using the Berlin Questionnaire. The Berlin Questionnaire consists of three categories designed to elicit information regarding snoring (category 1), daytime somnolence (category 2), and the presence of obesity and/or hypertension (category 3). Categories 1 and 2 are considered positive if 2 or more responses are positive category 3 is considered positive if 1 response is positive and/or the body mass index is greater than 30 kg per meter squared. A patient is considered to have a high likelihood of sleep disordered breathing if 2 or more categories are positive
Perceived social support | 16-24 weeks gestation
  Using the Multidimensional Scale of Perceived Social Support (MSPSS). MSPSS is a 12-item scale that measures the adequacy of social support. It consists of 3 subgroups that include items about family, friends and social support from a special person. It consists of 4 items for each group and each item is graded on a 7-item likert scale. A high total score indicates a high level of perceived social support.

CONTACTS AND LOCATIONS:
Overall Officials: Denice Feig, Principal Investigator — Lunenfeld-Tanenbaum Research Institute, Mount Sinai Hospital
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No